CLINICAL TRIAL: NCT01898039
Title: Allogeneic Vaccine Modified to Express HLA A2/4-1BB Ligand for High Risk or Low Residual Disease Melanoma Patients - Phase I/II Study.
Brief Title: Modified Vaccine for High Risk or Low Residual Melanoma Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0419-12-HMO-CTIL
Record Dates: First submitted 2013-05-09; First posted 2013-07-12 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-03

CONDITIONS: Malignant Melanoma
Keywords: malignant melanoma; vaccine; cell line; high risk; residual disease
MeSH Terms: conditions — Melanoma; Neoplasm, Residual | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A2/4-1BBL melanoma vaccine (Experimental): On days 1 and 2 patients will be sensitized to DNP by topically applying 0.1 ml of 2% DNP dissolved in acetone-corn oil (Sigma) to the inner aspect of the arm.
  On day 10, intravenous low dose cyclophosphamide, 300 mg/m2, will be administered at the day care unit. On day 14 the appropriate dose of irradiated M20/A2B cells will be injected into three adjacent sites on the upper arm or thigh, avoiding limbs where lymph node dissection had been previously performed. Four additional doses of the vaccine will be administered at intervals of 21 days.
  Interventions: Biological: A2/4-1BBL melanoma vaccine; Procedure: DNP sensititzation; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: A2/4-1BBL melanoma vaccine — On days 14, 35, 56, 77 and 98 the appropriate dose of irradiated M20/A2B cells will be injected into three adjacent sites on the upper arm or thigh, avoiding limbs where lymph node dissection had been previously performed.
  Other Names: M20/A2B vaccine
Procedure: DNP sensititzation — Include brand names, serial numbers and code names, if applicable. Other names are used to improve search results on the ClinicalTrials.gov web site.
  On days 1 and 2 patients will be sensitized to DNP by topically applying 0.1 ml of 2% DNP dissolved in acetone-corn oil (Sigma) to the inner aspect of the arm.
Drug: Cyclophosphamide — On day 10, intravenous low dose cyclophosphamide, 300 mg/m2, will be administered.

SUMMARY:
This study is designed for patients who had malignant melanoma and, following tumor removal, are now free of disease, or have only very minor residual disease, and are at a very high risk of disease recurrence. These patients will be treated with the A2/4-1BBL melanoma vaccine, a compatible melanoma cell line that has been engineered to express a molecule termed 4-1BBL, which enhances the chances of the cell line to be recognized by the patient's immune system, and to induce its stimulation. The hypothesis that drives the study states that the immune response against the cell line will also be effective against the residual tumor that may still be present in the body.

ELIGIBILITY:
Inclusion Criteria:

1. Patients included in this protocol must carry one or more of the following tissue typing alleles: HLA-A2, -A24, -A33, -B35, -B49, -CW04/12(04/08). We estimate that 50% of melanoma patients will be eligible.
2. Cutaneous malignant melanoma AJCC stage IIb (>4 mm) or IIc (ulcerated melanoma >4mm).
3. Metastatic melanoma AJCC stage III (nodal involvement, N1-3a,b) post-surgical removal of lymph nodes.
4. Metastatic melanoma AJCC stage IV, completely resected.
5. Non-resectable metastatic melanoma of low burden disease and normal LDH who have undergone at least two treatment lines, including chemotherapy (DTIC, temodal, taxanes, platinum compounds), anti-CTLA-4 (ipilimumab) and B-RAF inhibitor if harboring the V600E BRAF mutation in their tumor.
6. Non cutaneous malignant melanoma of respective stages including uveal and mucosal melanoma.
7. Melanoma can be of either mutant or wild-type B-RAF.
8. Karnofsky performance status > 80 (Normal activity with effort).
9. No active cardio-respiratory disease.
10. Not pregnant or nursing. Women must take contraceptives during the treatment period.Hematocrit >25% and WBC >3000.
11. Informed consent of the patient.

Exclusion Criteria:

1. Administration of cytotoxic drugs or extensive radiotherapy less than 28 days prior to protocol administration.
2. Active brain metastases requiring corticosteroids.
3. Concurrent malignancy (other than skin cancer, carcinoma in situ of cervix and early stage prostate cancer).
4. Active serious infection.
5. Allergy to penicillin.
6. Patient's will to withdraw from the study at any stage.
7. HIV and chronic hepatitis B and C carrier

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-05; Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
grade 2-4 adverse events according to CTCEA criteria | Day 1
monitoring anti-tumor immune response | Day 0
  Anti-tumor immune response will be measured by delayed type hypersensitivity in vivo and by in vitro lymphocyte response.
grade 2-4 adverse events according to CTCEA criteria | Day 28
grade 2-4 adverse events according to CTCEA criteria | Day 56
grade 2-4 adverse events according to CTCEA criteria | month 3
grade 2-4 adverse events according to CTCEA criteria | month 4
grade 2-4 adverse events according to CTCEA criteria | month 5
grade 2-4 adverse events according to CTCEA criteria | month 6
monitoring anti-tumor immune response | Day 28
  Anti-tumor immune response will be measured by delayed type hypersensitivity in vivo and by in vitro lymphocyte response
monitoring anti-tumor immune response | Day 56
  Anti-tumor immune response will be measured by delayed type hypersensitivity in vivo and by in vitro lymphocyte response
monitoring anti-tumor immune response | month 3
  Anti-tumor immune response will be measured by delayed type hypersensitivity in vivo and by in vitro lymphocyte response
monitoring anti-tumor immune response | month 4
  Anti-tumor immune response will be measured by delayed type hypersensitivity in vivo and by in vitro lymphocyte response
monitoring anti-tumor immune response | month 5
  Anti-tumor immune response will be measured by delayed type hypersensitivity in vivo and by in vitro lymphocyte response
monitoring anti-tumor immune response | month 6
  Anti-tumor immune response will be measured by delayed type hypersensitivity in vivo and by in vitro lymphocyte response

SECONDARY OUTCOMES:
overall survival and disease free survival | D1, Mo6, Mo10, Mo14, Mo18, Mo20, Mo24 and every 4 months till year 5

CONTACTS AND LOCATIONS:
Locations (1):
- Sharett Institute of Oncology, Hadassah Medical Organization, Jerusalem, Israel